CLINICAL TRIAL: NCT04605861
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Phase III Trial to Evaluate the Efficacy and Safety of Liraglutide on Body Weight Loss in Obese and Overweight Patients
Brief Title: The Efficacy and Safety of Liraglutide on Body Weight Loss in Obese and Overweight Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JSWB-LRG2020-301
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Obese; Overweight
Keywords: weight loss; obeses; overwweight; Liraglutide
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical trial. The total study duration is 34~36 weeks, including 2-week screening, 6~8-week dosage titration, 24-week stable treatment and 2-week safety follow-up.
Who Masked: Participant, Investigator
Masking Description: Regardless of treatment allocations, each subject receive the same total volume of investigational drug or placebo. All drug automatic injectors and kits, study drugs or placebo are identical in appearance and labels to blind subjects and investigators. This can minimize the bias of investigators and subjects on treatment evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide Injection, once a day, injected subcutaneously on abdomen, thigh or upper arm.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo (Liraglutide Injection simulator), once a day, injected subcutaneously on abdomen, thigh or upper arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Liraglutide Injection, once a day, injected subcutaneously on the sites of abdomen, thigh or upper arm. The initial dose of Liraglutide Injection will be 0.6 mg per day. The dose is escalated every one to two weeks to reduce the gastrointestinal symptoms. At Week 7, the dose is increased to 3.0 mg per day. For the subjects who are not able to tolerate the target dose of 3.0 mg,the dose is reduced to 2.4 mg a day and escalated to the dose to 3.0 mg within two weeks. If the subjects are still unable to tolerate this dose (3.0 mg), the treatment is terminated.
  Arms: Liraglutide
Drug: Placebo — Placebo Injection, once a day, injected subcutaneously on the sites of abdomen, thigh or upper arm. The initial dose of Placebo Injection will be 0.6 mg per day. The dose is escalated every one to two weeks to reduce the gastrointestinal symptoms. At Week 7, the dose is increased to 3.0 mg per day. For the subjects who are not able to tolerate the target dose of 3.0 mg,the dose is reduced to 2.4 mg a day and escalated to the dose to 3.0 mg within two weeks. If the subjects are still unable to tolerate this dose (3.0 mg), the treatment is terminated.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo controlled trial to evaluate the effect and safety of Liraglutide Injection on body weight loss compared with placebo in obese or overweight adult patients with comorbidity of metabolic disorders.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical trial. The total study duration is 34~36 weeks, including 2-week screening period, 6~8-week dosage titration, 24-week stable treatment and 2-week safety follow-up period. Subjects with obesity or overweight with comorbidity of metabolic disorders receive subcutaneous injection of 3.0 mg Liraglutide or placebo every day. The primary endpoint is the change of body weight or the percentage of body weight loss greater than 5%. The changes of body weight between Liraglutide Injection group and placebo group will be compared. In the course of the trial, the subjects are weighted on fasting state. Blood samples are collected according to the protocol. All subjects receive lifestyle intervention, including a reductiong of calorie intake by 500 kcal a day and physical exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Those voluntarily participating and signing the ICF.
2. Those aged 18-70 years old (including 18 and 70 years old), without restriction on male and female
3. Those failing to control their body weight in previous diet therapy alone.
4. Those voluntarily following the medication, diet and exercise requirements decided by the investigators.
5. Those with a stable body weight (patient reported body weight change < 5 kg) in last 3 months.
6. Those with BMI ≥ 30 kg/m2 (obese) or BMI ≥ 27 kg/m2 (overweight) accompanied by at least one treated or untreated related metabolic abnormality (hypertension, dyslipidemia, type 2 diabetes). Those with untreated hypertension defined as SBP ≥ 140 mmHg or DBP ≥ 90 mmHg; untreated dyslipidemia defined as LDL-C ≥ 4.1 mmol/L, TG ≥ 1.7 mmol/L, TC ≥ 5.7 mmol/L or HDL-C < 1.0 mmol/L in male and < 1.3 mmol/L in female.
7. Those with type 2 diabetes should additionally meet the following inclusion criteria:

   1. Those diagnosed as type 2 diabetes according to WHO (1999) Diagnostic and Classification Criteria at the time of screening;
   2. Those receiving diet and exercise therapy alone, or receivig metformin, sulfonylureas, glycosidase inhibitors and glinides alone or in combination on the basis of diet and exercise therapy, with their treatment remaining stable at least 3 months before screening (with original documents such as prescriptions provided);
   3. Those with HbA1c of 7.0-10.0% (inclusive);
   4. Those with FPG < 13.3 mmol/L (240 mg/dL).

Exclusion Criteria:

Subjects who meet one of the following exclusion criteria will be excluded.

1. Those with type 1 diabetes or secondary diabetes.
2. Those with acute metabolic complications such as diabetic ketoacidosis or hyperglycemia (coma) within 6 months before screening.
3. Those with 2 or more severe hypoglycemia events (hypoglycemia with severe cognitive impairment and need other measures to help them recover) without obvious inducement within 3 months before screening.
4. Those receiving GLP-1 receptor agonist, DPP-4 inhibitors, SGLT-2 inhibitor, or insulin therapy within 3 months prior to screening.
5. Those with obesity caused by endocrine diseases such as Cushing's syndrome.
6. Patients taking drugs that can significantly increase weight in the 3 months before screening, including systemic glucocorticoid (except cumulative or continuous use of less than 14 days).
7. Those using OTC weight-loss drugs or appetite inhibitors (including traditional Chinese medicine as weight-loss drugs) within 1 month before screening, or use prescription weight-loss drugs (such as fentanyl, sibutramine, orlistat) or lipid dissolving injection (such as fat dissolving needle) within 3 months before screening.
8. Those with binge eating behavior in the past, that is, eating a large amount of food in a short period of time with a sense of loss of control.
9. Those who have treated or plan to treat obesity (during the trial) with surgery or body weight loss devices.
10. Those with a past or family history of MTC (grandparents, parents, siblings), or those whose genetic diseases are prone to induce MTC and MEN2.
11. Those with thyroid nodules of unknown etiology at the time of screening which is considered clinically significant by the investigator (calcitonin is more than 50 pg/ml, which is only allowed to be retested once).
12. Those with a past history or found to have hyperthyroidism or hypothyroidism or subclinical hypothyroidism at the time of screening [TSH > 6 mIU/L].
13. Those with history of pancreatic cancer, acute or chronic pancreatitis, or with acute or chronic pancreatitis at the time of screening, or having blood amylase or lipase ≥ 3 times ULN.
14. Those with acute gallbladder disease (cholecystitis, gallstone) more than 2 times in 1 year before screening.
15. Those with MDD, anxiety disorder or other mental illnesses or with the PHQ-9 score ≥ 15 at screening
16. Those with the following cardiovascular and cerebrovascular diseases within 6 months before screening: decompensated cardiac insufficiency (NYHA Class III-IV), UA or AMI, CVA or stroke.
17. Those with a history of heart valve replacement, CABG or other PTCA including percutaneous coronary intervention.
18. Those who fail to control their blood pressure effectively, with SBP ≥ 160 mmHg or DBP ≥ 100 mmHg.
19. Those with a history of malignancy in the past 5 years, not including cervical epithelial carcinoma, squamous cell carcinoma or basal cell carcinoma of skin that have been clinically cured within 5 years.
20. Those with known proliferative retinopathy or maculopathy.
21. Those with a history of major surgical operations (intrathoracic, intracranial, intraperitoneal, etc.) within 6 months, or planning to perform operations that may interfere with the completion or compliance of the study.
22. Those with a history of organ transplantation.
23. Those with ADIS or syphilis at the time of screening, or whose serum virological test shows hepatitis C virus antibody or hepatitis B surface antigen and hepatitis B core antibody are positive at the time of screening.
24. Those with AST or ALT > 3.0-fold ULN, or total bilirubin > 2.0-fold ULN at the time of screening.
25. Those with eGFR < 60 mL/min/1.73 m2 at the time of screening.
26. Those with a history of drug abuse (heavy and repeated use of dependent drugs or substances not related to medical purposes, including addictive and habitual drugs, causing physical and mental dependence) in 5 years before screening and alcohol dependence (long-term heavy drinking, causing physical and mental dependence, male drinking more than 14 units of alcohol per week, and female drinking more than 7 units per week) (1 unit alcohol = 360 mL beer or 45 mL spirits with 40% alcohol content or 150 mL wine)].
27. Female who are known to be pregnant (determined by pregnancy test at the time of screening) or who are breast-feeding or who plan a pregnancy during the study and are unwilling to take effective contraceptive measures (including partners).
28. Those participating in other intervention clinical trials within 3 months prior to screening.
29. Those known to be allergic to GLP-1 receptor agonist.
30. Those with any serious systemic diseases as determined by the investigator, or other diseases as believed by the investigator to be possible to interfere with the results of this study or abnormal laboratory tests with clinical significance.
31. Those who, according to the opinion of investigators, are not suitable to participate in clinical trials, including those who are physically or psychologically unable to comply with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
The percentage of body weight loss | through study completion, an average of 32 weeks
  The percentage of body weight loss from baseline to the end of treatment
The proportion of body weight loss ≥ 5 percent | through study completion, an average of 32 weeks
  The proportion of subjects whose body weight loss is greater than ≥ 5 percent from baseline level to the end of treatment

SECONDARY OUTCOMES:
Changes in waist circumference | through study completion, an average of 32 weeks
  Changes in waist circumference of the subjects at the end of treatment
Changes in diastolic pressure and systolic pressure | through study completion, an average of 32 weeks
  Changes in blood pressure level (diastolic pressure and systolic pressure) of the subjects at the end of treatment
Changes in pulse of the subjects | through study completion, an average of 32 weeks
  Changes in pulse of the subjects at the end of treatment
The changes in blood lipid | through study completion, an average of 32 weeks
  The changes in blood lipid levels (triglyceride, total cholesterol, low density lipoprotein cholesterol, and high density lipoprotein cholesterol) of the subjects at the end of treatment
The changes in blood glucose | through study completion, an average of 32 weeks
  The change in fasting blood-glucose of the subjects at the end of treatment
The changes in HbA1c | through study completion, an average of 32 weeks
  The changes in HbA1c of patients with type 2 diabetes at the end of treatment
Absolute body weight change | through study completion, an average of 32 weeks
  The absolute body weight loss of the subjects at the end of treatment
The proportion of body weight loss > 10 percent | through study completion, an average of 32 weeks
  The proportion of subjects with body weight loss > 10 percent at the end of treatment
The changes in IWQOL-lite | through study completion, an average of 32 weeks
  Effect of changes in body weight of the patients to the IWQOL-lite at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hosital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT04605861/Prot_SAP_000.pdf